## INFORMED CONSENT TERM (2 copies)

| I, | RG | | agree to |
|---|---|---|---|
| participate and authorize n | nv inclusion in | the study | "EFFECT OF |
| DEXAMETHASONE, ONDANSET | | | |
| RECOVERY AFTER THE ADMI | NISTRATION OF I | NTRATECAL I | MORPHINE IN |
| PATIENTS SUBMITTED TO S | URGICAL CORREC | TION OF FR | RACTURES OF |
| INFERIOR MEMBERS". The aim | | | |
| quality of anesthesia recovery in | - | | |
| (anti-inflammatory) or ondanse | | | |
| already used in other surgeries p | _ | | |
| know if it would also be helpfu | | | |
| which is the anesthetic propose | | | |
| name will remain confidential an | | | |
| clarified that I will not have any<br>aware that I may suspend my c | | , . | |
| prejudice to my treatment of the | - | - | - |
| occur should be referred to | | | |
| Department of Anesthesiology of | | - | |
| Sorocaba (CCMB / PUC-SP), telep | | | |
| , | () ( | | |
| Sorocaba, | of | | |
| (name of volunteer) (signatur | re of volunteer) | | |
| (name of witness) (signature | of witness) | | |
| manie or withess) (signature | or withtess; | | |
| (researcher's name) (research | ner's signature) | | |